CLINICAL TRIAL: NCT01772316
Title: A Multicenter, Open-label, Long-term Extension Study of WA22762 and NA25220 to Evaluate Safety and Efficacy of Subcutaneous Tocilizumab in Patients With Moderate to Severe Rheumatoid Arthritis
Brief Title: A Long-Term Extension Study of WA22763 and NA25220 of Subcutaneous RoActemra/Actemra (Tocilizumab) in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28488; 2012-002632-87 (EudraCT Number)
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tocilizumab Subcutaneous (SC) (Experimental): Participants received Tocilizumab 162 milligram (mg) given as 0.9 milliliter (mL) of a 180 milligram per milliliter (mg/mL) solution administered once a week (for participants entering from NCT01194414) or once every two weeks (for participants entering from NCT01232569) by SC injection and as a single fixed dose irrespective of body weight.
  Interventions: Drug: tocilizumab

INTERVENTIONS:
Drug: tocilizumab — 162 mg subcutaneously weekly or every two weeks, 96 weeks
  Other Names: Roactemra

SUMMARY:
This multicenter, open-label, single arm, long-term extension study will evaluate the safety and efficacy of RoActemra/Actemra (tocilizumab) in participants with moderate to severe rheumatoid arthritis who have completed the 97-week WA22762 or the 96-week NA25220 core study. Participants will receive RoActemra/Actemra 162 milligram (mg) subcutaneously weekly (for participants entering from WA22762) or every two weeks (for participants entering from NA25220) for 96 weeks, with telephone call follow-up visits at Weeks 100 and 104.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Participants who have completed the 97-week WA22762 or 96-week NA25220 core study on subcutaneous or intravenous RoActemra/Actemra and based on the investigator's judgment may continue to benefit from RoActemra/Actemra treatment in this study investigating the subcutaneous formulation
* Oral corticosteroids and non-steroidal anti-inflammatory drugs (NSAIDS) up to the maximum recommended dose are permitted if on a stable dose regimen for >/= 4 weeks prior to baseline
* Permitted non-biological disease-modifying anti-rheumatic drugs (DMARDs) are allowed
* Receiving treatment on an outpatient basis
* Females of childbearing potential and males with female partners of childbearing potential must agree to use reliable means of contraception

Exclusion Criteria:

* Participants who have prematurely withdrawn from the WA22762 or NA25220 core studies for any reason
* Previous treatment with any cell-depleting therapies, including investigational agents or approved therapies
* History of severe allergic or anaphylactic reactions to human, humanized or mural monoclonal antibodies
* Evidence of serious uncontrolled concomitant disease
* Current liver disease as determined by the principal investigator
* History of diverticulitis, diverticulosis requiring antibiotic treatment or chronic ulcerative lower gastrointestinal (GI) disease such as Crohn's disease, ulcerative colitis or other symptomatic lower GI conditions that might predispose to perforations
* Known active current or history of recurrent infections
* Any major episode of infection requiring hospitalization or treatment with intravenous (IV) antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Active tuberculosis requiring treatment within the previous 3 years
* Primary or secondary immunodeficiency (history of or currently active)
* Pregnant or breast feeding women
* Body weight > 150 kilogram (kg)
* Inadequate renal, hepatic or hematologic function
* Positive for hepatitis B or hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Spain (11):
  - Mérida, Badajoz
  - Santander, Cantabria
  - A Coruña, La Coruña
  - Santiago de Compostela, La Coruña
  - Madrid, Madrid
  - Málaga, Malaga
  - Seville, Sevilla
  - San Cristóbal de La Laguna, Tenerife
  - Valenica, Valencia
  - Barakaldo, Vizcaya
  - Bilbao, Vizcaya

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 47 participants were enrolled in the trial and received treatment. All participants enrolled were included in the safety analysis. Of the 47 participants, 13 participants were not included in the statistical analysis for outcome measures because they did not meet eligibility criteria.
Groups:
- Tocilizumab Subcutaneous (SC): Participants received Tocilizumab 162 milligram (mg) given as 0.9 milliliter (mL) of a 180 milligram per milliliter (mg/mL) solution administered once a week (for participants entering from NCT01194414) or once every two weeks (for participants entering from NCT01232569) by subcutaneous (SC) injection and as a single fixed dose irrespective of body weight.
Period: Overall Study
Arm/Group | Tocilizumab Subcutaneous (SC)
Started | 47
Completed | 40
Not Completed | 7
Not completed — Serious adverse event | 1
Not completed — Inform consent withdrawn | 1
Not completed — Withdrawn by sponsor decision | 5

BASELINE CHARACTERISTICS:
Groups:
- Tocilizumab Subcutaneous (SC): Participants received Tocilizumab 162 mg given as 0.9 mL of a 180 mg/mL solution administered once a week (for participants entering from NCT01194414) or once every two weeks (for participants entering from NCT01232569) by SC injection and as a single fixed dose irrespective of body weight.
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant that was administered study drug, regardless of causal attribution.
Time Frame: Baseline up to follow-up (Week 104)
Population: All participants receiving study drug were included in the safety analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 47
percentage of participants | 83

2. Primary Outcome: Percentage of Participants Withdrawn From the Study Due to Lack of Therapeutic Response
Time Frame: Baseline up to follow-up (Week 104)
Population: Per-protocol population included all participants who had at least one dose of study medication and at least one safety evaluation after dose administration.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 34
percentage of participants | 0

3. Primary Outcome: Change From Baseline in Disease Activity Score 28 - Erythrocyte Sedimentation Rate (DAS28-ESR) at Week 48
Description: The DAS28 is a combined index for measuring disease activity in rheumatoid arthritis. The index included swollen joint count (SJC), tender joint count (TJC), acute phase response (ESR or high sensitivity C-reactive protein [hsCRP]) and general health status (GH). For this study, ESR was used to calculate DAS28 score. The index was calculated using the following formula: DAS28 = (0.56 × √[TJC 28]) + (0.28 × √[SJC 28]) + (0.7 × ln[ESR]) + (0.014 × GH). The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. Change in DAS28ESR=DAS28-ESR at Week 48 - DAS28-ESR at Baseline.
Time Frame: Baseline, Week 48
Population: Per-protocol population included all participants who had at least one dose of study medication and at least one safety evaluation after dose administration. Number of participants analyzed represent number of participants who were evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 30
units on a scale
  Baseline | 2.9 (1.4)
  Change at Week 48 | -0.832 (0.292)

4. Primary Outcome: Change From Baseline in DAS28-ESR at Week 96
Description: The DAS28 is a combined index for measuring disease activity in rheumatoid arthritis. The index included SJC, TJC, acute phase response (ESR or high sensitivity C-reactive protein [hsCRP]) and general health status. For this study, ESR was used to calculate DAS28 score. The index was calculated using the following formula: DAS28 = (0.56 × √[TJC28]) + (0.28 × √[SJC28]) + (0.7 × ln[ESR]) + (0.014 × GH). The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. Change in DAS28ESR=DAS28-ESR at Week 96 - DAS28-ESR at Baseline.
Time Frame: Baseline, Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 30
units on a scale | -0.804 (0.230)

5. Primary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Week 48
Description: The SDAI was the numerical sum of five outcome parameter: SJC and TJC, Patient Global Assessment of Disease Activity (PGA) and Investigator Global Assessment of Disease Activity (IGA), and level of hsCRP. The index was calculated using the following formula SDAI = TJC28 + SJC28 + PGA + IGA + CRP. Change in SDAI = SDAI at Week 48 - SDAI at Baseline. SDAI total score = 0-86. SDAI <=3.3 indicates clinical remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high (or severe) disease activity. Here, n signifies the number of subjects evaluable at the specified time points.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 30
units on a scale
  Baseline | 12.2 (10.7)
  Change at Week 48 | -7.572 (2.115)

6. Primary Outcome: Change From Baseline in SDAI at Week 96
Description: The SDAI was the numerical sum of five outcome parameter: SJC and TJC, PGA and IGA, and level of hsCRP. The index was calculated using the following formula SDAI = TJC28 + SJC28 + PGA + IGA + CRP. Change in SDAI = SDAI at Week 96 - SDAI at Baseline. SDAI total score = 0-86. SDAI <=3.3 indicates clinical remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high (or severe) disease activity.
Time Frame: Baseline, Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 30
units on a scale | -6.599 (2.210)

7. Primary Outcome: Change From Baseline in Total Tender Joint Count (TJC) at Week 48
Description: An assessment of 66 joints for swelling and 68 joints for tenderness was made. Joints were assessed and classified as tender/not tender and swollen/not swollen by pressure and joint manipulation on physical examination. A smaller number indicated improvement. Here, 'n' represents the number of participants with a measure at specified time point.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 33
units on a scale
  Baseline | 2.5 (4.1)
  Change at Week 48 | 1.3 (2.0)

8. Primary Outcome: Change From Baseline in Total TJC at Week 96
Description: An assessment of 66 joints for swelling and 68 joints for tenderness was made. Joints were assessed and classified as tender/not tender and swollen/not swollen by pressure and joint manipulation on physical examination. A smaller number indicated improvement.
Time Frame: Baseline, Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 33
units on a scale | 1.5 (3.6)

9. Primary Outcome: Change From Baseline in Swollen Joint Count (SJC) at Week 48
Description: An assessment of 66 joints for swelling and 68 joints for tenderness was made. Joints were assessed and classified as tender/not tender and swollen/not swollen by pressure and joint manipulation on physical examination. A negative number indicated improvement.
Time Frame: Baseline, Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 34
units on a scale
  Baseline | 1.8 (3.4)
  Change at Week 48 | -1.531 (0.587)

10. Primary Outcome: Change From Baseline in SJC at Week 96
Description: An assessment of 66 joints for swelling and 68 joints for tenderness was made. Joints were assessed and classified as tender/not tender and swollen/not swollen by pressure and joint manipulation on physical examination. Change in SJC = SJC at Week 96 - SJC at Baseline. A negative number indicated improvement.
Time Frame: Baseline, Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 34
units on a scale | -1.188 (0.543)

11. Secondary Outcome: Percentage of Participants With Remission (DAS28 <2.6 or SDAI </=3.3) at Weeks 48 and 96
Time Frame: Week 48, Week 96
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 34
percentage of participants
  DAS <2.6 at Week 48 | 71.9
  DAS <2.6 at Week 96 | 62.5
  SDAI </=3.3 at Week 48 | 28.6
  SDAI </=3.3 at Week 96 | 29.6

12. Secondary Outcome: Percentage of Participants With Disease-Modifying Antirheumatic Drugs (DMARDs)/Corticosteroid Dose Reductions and/or Discontinuation
Time Frame: Randomization of first participant to clinical cutoff date (19MAY2015) (approximately 29 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 34
percentage of participants | 38.2

13. Secondary Outcome: Patient Global Visual Analog Score (VAS) at Specified Time Points
Description: This assessment represents the patient's overall assessment of their current disease activity on a 100 millimeter (mm) horizontal VAS. The extreme left end of the line should be described as "no disease activity" (symptom free and no arthritis symptoms) and the extreme right end as "maximum disease activity" (maximum arthritis disease activity). Scores ranged from 0 to 100 with a higher score indicating more disease activity. A negative change score indicated less disease activity.
Time Frame: Baseline, Week 48, Week 96
Population: Per-protocol population included all participants who had at least one dose of study medication and at least one safety evaluation after dose administration. Here, 'n' represents the number of participants with a measure at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 34
units on a scale
  Baseline (n=34) | 30.8 (21.8)
  Week 48 (n=33) | 30.0 (22.6)
  Week 96 (n=33) | 26.0 (21.8)

14. Secondary Outcome: Patient Pain VAS Score at Specified Time Points
Description: This assessment represents the patient's assessment of his/her current level of pain on a 100 mm horizontal VAS. The extreme left end of the line should be described as "no pain" and the extreme right end as "unbearable pain". Scores ranged from 0 to 100 with a higher score indicating more pain. A negative change score indicated less pain.
Time Frame: Baseline, Week 48, Week 96
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 34
units on a scale
  Baseline (n=34) | 32.4 (21.8)
  Week 48 (n=33) | 29.8 (21.3)
  Week 96 (n=33) | 27.0 (22.2)

15. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Specified Time Points
Description: The HAQ-DI is a questionnaire specific for rheumatoid arthritis and consists of 20 questions referring to 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Minimum score was 0, maximum score was 3. A smaller score indicated improvement.
Time Frame: Baseline, Week 48, Week 96
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Subcutaneous (SC)
Number analyzed (Participants) | 34
units on a scale
  Baseline (n=34) | 0.8 (0.6)
  Week 48 (n=33) | 0.7 (0.5)
  Week 96 (n=33) | 0.8 (0.7)

ADVERSE EVENTS:
Time Frame: Baseline up to follow-up (Week 104)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant that was administered study drug, regardless of causal attribution.
Arm/Group | Tocilizumab Subcutaneous (SC)
Serious Adverse Events (participants affected / at risk) | 3/47
Other Adverse Events (participants affected / at risk) | 39/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Subcutaneous (SC) (N=47)
Renal colic (Renal and urinary disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Subcutaneous (SC) (N=47)
Neutropenia (Blood and lymphatic system disorders) | 3
Gastroenteritis (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 13
Urinary tract infection (Infections and infestations) | 5
Wound (Injury, poisoning and procedural complications) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.